CLINICAL TRIAL: NCT01211535
Title: Subjective Comfort With Multipurpose Care Solutions in Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMA-09-59
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-10

CONDITIONS: Myopia; Astigmatism; Refractive Error
Keywords: Soft contact lenses; Multi-purpose Solution
MeSH Terms: conditions — Myopia; Astigmatism; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTI-FREE RepleniSH (Experimental): OPTI-FREE RepleniSH multipurpose solution used with study contact lenses on a daily wear basis for 14 days
  Interventions: Device: OPTI-FREE RepleniSH multipurpose solution; Device: Silicone hydrogel contact lenses
- ReNu Biotrue (Active Comparator): ReNu Biotrue multipurpose solution used with study contact lenses on a daily wear basis for 14 days
  Interventions: Device: ReNu Biotrue multipurpose solution; Device: Silicone hydrogel contact lenses

INTERVENTIONS:
Device: OPTI-FREE RepleniSH multipurpose solution — FDA-approved, multipurpose solution used as indicated for cleaning, rinsing, conditioning, disinfecting, and storing study contact lenses on a daily wear basis for 14 days
  Other Names: OPTI-FREE® RepleniSH®
  Arms: OPTI-FREE RepleniSH
Device: ReNu Biotrue multipurpose solution — FDA-approved, multipurpose solution used as indicated for cleaning, disinfecting, daily protein removing, and storing study contact lenses on a daily wear basis for 14 days
  Other Names: ReNu Biotrue™
  Arms: ReNu Biotrue
Device: Silicone hydrogel contact lenses — Silicone hydrogel contact lenses per subject's habitual brand and prescription worn on a daily wear basis for 14 days, with either OPTI-FREE RepleniSH or ReNu Biotrue used for contact lens care

SUMMARY:
The purpose of this study was to assess the comfort of OPTI-FREE RepleniSH in soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing silicone hydrogel contact lenses on a daily wear basis;
* Currently using OPTI-FREE RepleniSH contact lens solution;
* Generally healthy;
* Normal ocular health;
* Willing to follow study procedures and visit schedule;
* Sign Informed Consent and privacy document;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of additional lens cleaners;
* Known sensitivities to any ingredient in either test article;
* Systemic or ocular disease or disorder that would negatively affect the conduct or outcome of the study;
* History of ocular surgery/trauma within the last 6 months;
* Any topical ocular or systemic antibiotics within 7 days of enrollment continuing throughout the study;
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollent;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Trial Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPTI-FREE RepleniSH | ReNu Biotrue
Started | 52 | 52
Completed | 52 | 51
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPTI-FREE RepleniSH | ReNu Biotrue | Total
Number analyzed (Participants) | 52 | 52 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.4) | 35.4 (10.96) | 34.3 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 0) in Ocular Comfort Rating at Day 14
Description: Ocular comfort was rated by the participant on a continuous visual analog scale from 0-100, where 0=extremely uncomfortable, 50=neither comfortable nor uncomfortable, and 100=extremely comfortable. The participant marked a horizontal line across the scale at the point that best described, "how your eyes feel right now." A positive number indicates increased ocular comfort; a negative number indicates decreased ocular comfort.
Time Frame: Baseline (Day 0), Day 14
Population: All participants who received regimen, satisfied inclusion/exclusion criteria, and completed the 14-day treatment period (per protocol)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | OPTI-FREE RepleniSH | ReNu Biotrue
Number analyzed (Participants) | 52 | 51
Units on a scale
  Baseline (Day 0) | 87.40 [83.82 to 90.99] | 88.79 [85.21 to 92.37]
  Day 14 | 81.75 [78.17 to 85.33] | 83.18 [79.56 to 86.79]
  Change from Baseline (Day 0) at Day 14 | -5.65 [-10.72 to -0.59] | -5.61 [-10.70 to -0.52]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: The safety population includes all participants who received study regimen.
Arm/Group | OPTI-FREE RepleniSH | ReNu Biotrue
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other